CLINICAL TRIAL: NCT03366909
Title: Mindfulness Meditation and Cannabis Dependence : Therapy Effectiveness
Acronym: MACBETH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-A01466-47
Record Dates: First submitted 2017-11-23; First posted 2017-12-08 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Addiction; Cannabis Use; Cannabis Dependence
Keywords: mindfulness; cannabis use
MeSH Terms: conditions — Behavior, Addictive; Marijuana Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBRP group (Experimental): 20 patients 2 groups of 10 patients
  Interventions: Behavioral: Mindfulness based relapse prevention (MBRP)
- classic care in addictology center (Active Comparator): 20 patients
  Interventions: Behavioral: classic therapy

INTERVENTIONS:
Behavioral: Mindfulness based relapse prevention (MBRP) — These weekly visits include a Mindfulness Meditation session:
  The sessions of meditation take place in a dedicated room. The collective sessions owed approximately of 2 hours and will approach the following themes: (1) Autopilot, (2) Facing obstacles, (3) Full awareness of breath, (4) Staying present, (5) Allow, let go (6) Thoughts are not facts, (7) How to take care of oneself, (8) Mindfulness on a daily basis.
  Arms: MBRP group
Behavioral: classic therapy — These weekly visits include usual addiction care provided during a consultation. This care includes psychotherapeutic management: brief interventions, cognitive-behavioral therapies, motivational interviews; associated with nonsystematic pharmacological management.
  Arms: classic care in addictology center

SUMMARY:
Cannabis use can lead to addiction in about 5 to 10 % of users in France. Currently, behavioral interventions are the most dependable but effectiveness is still reduced. Mindfulness meditation has demonstrated an effectiveness in several meta analysis (anxiety and depressive disorder) and seems to be relevant to reduce anxious and impulsive symptoms found in cannabis use disorders.

This study proposes to determinate the mindfulness effectiveness in reduction of cannabis use in regular consumer. The consumption decrease is estimated with a retrospective diary, TLFB (Timeline Follow Back) which collect cannabis use every week until the 12th. Urine (week 0/baseline, 2, 4, 6, 8, 10, 12) and hair (week 0/baseline, 10) analyses are regularly effected.

Patients included in control group get classic cares in an addictology center in CHRU of Nancy. Patients included in mindfulness group receive one session a week during eight weeks (MBRP protocol : Mindfulness -Based Relapse Prevention). The study process goes on for 12 weeks.

An ancillary study measures the impact of cannabis decreases on retinal electrophysiological and architectural markers, usually disturbed by cannabis uses.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 55
* cannabis use: more than 7 joint a week or diagnostic of abuse/dependence at MINI (mini international neuropsychiatric interview)
* Recent use authenticated in urine
* patient voluntary to stop cannabis use
* patient with social security
* written consent for study

Exclusion Criteria:

* alcohol dependence (AUDIT: alcohol use disorders test)
* other psychoactive substance abuse or dependence (DSM 4)
* Progressive psychiatric disorder (MINII) excepted anxious disorder)
* Current neurologic disorder
* Patient deficiency with difficulty or impossibility to understand informations
* protection of vulnerable adults as guardianship or judicial protection
* pregnant or breastfeeding woman
* vital emergency
* no social security
* participation in another interventional study
* current retinal disorder (ancillary study)
* chronic glaucoma (ancillary study)
* opthalmologic disease decreasing visual acuity (ancillary study)
* current ocular infection

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2019-08-30 (Estimated); Study Completion 2020-02-27 (Estimated)

PRIMARY OUTCOMES:
Change in cannabis use between the baseline and the 8th week of treatment | At baseline, weeks 7 and 8
  The number of days of cannabis use (addition weeks 7 and 8) will be compared to the " less than or equal to 4 days"target.

SECONDARY OUTCOMES:
Number of patients who stopped cannabis 2 weeks after 8 weeks of treatment | at week 10
  measured by the absence of THC and metabolites in urinary and hair samples and the absence of cannabis use mentioned in the Timeline Follow Back retrospective diary (TLFB)
Patient retention rate at the end of treatment | at week 8
  number of patients who continue study until week 8
Severity of withdrawal symptoms questionnaire | At week 2, 4, 6, 8, 10, 12
  measured by the Cannabis Withdrawal Scale (CWS)
ERG : electroretinogram. | week 0, 8, 12
  measures a and b on ERG flash Measures P50 and N95 on ERG pattern
Thickness of retinal structure | at week 0 and 12
  measured by Optical Coherence Tomography (OCT)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Laprevote, Principal Investigator — Centre Psychothérapique de Nancy

IPD SHARING:
Plan to Share IPD: No